CLINICAL TRIAL: NCT05641363
Title: Comparison of Ketorolac at Three Doses in Children With Acute Pain: A Randomized Controlled Trial
Brief Title: Comparison of Ketorolac at Three Doses in Children With Acute Pain
Acronym: KETODOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Mohamed Eltorki, MBChB, Assistant Professor, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KETODOSE20221107
Record Dates: First submitted 2022-11-07; First posted 2022-12-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain; Abdominal Pain; Migraine; Appendicitis Acute; Renal Colic; Biliary Colic
MeSH Terms: conditions — Acute Pain; Abdominal Pain; Migraine Disorders; Appendicitis; Renal Colic | interventions — Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double dummy design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard dose group A (Active Comparator): IV ketorolac 0.5 mg/kg/dose up to a maximum dose of 30 mg plus IV normal saline placebo given at 0.25 mg/kg to a maximum of 30 mg plus IV normal saline placebo given at 0.5 mg/kg to a maximum of 10 mg
  Interventions: Drug: Ketorolac Tromethamine
- Low dose group B1 (Experimental): IV ketorolac 0.5 mg/kg to a maximum of 10 mg plus IV normal saline placebo given at 0.25 mg/kg to a maximum of 30 mg plus IV normal saline placebo given at 0.5 mg/kg to a maximum of 30 mg
  Interventions: Drug: Ketorolac Tromethamine
- Low dose group B2 (Experimental): IV ketorolac 0.25 mg/kg to a maximum of 30 mg plus IV normal saline placebo given at 0.5 mg/kg to a maximum of 30 mg plus IV normal saline placebo 0.5 mg/kg to a maximum of 10 mg
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — ketorolac tromethamine, an NSAID belonging to a group of non-opioid analgesics that inhibit the synthesis of prostaglandins and thromboxanes with strong analgesic and anti-inflammatory properties. It is the only non-opioid parenteral non-sedating analgesic available for use to treat acute pain in the emergency department.
  Other Names: ketorolac; toradol; intravenous ketorolac

SUMMARY:
Hospital Scene #1: A 6-year-old arrives in the Emergency Department at McMaster Children's Hospital (MCH) complaining of pain in his lower right side. His Dad explains the pain has been going on for a few hours and that Advil and Tyelnol haven't helped at all. He's anxious and concerned about his son because he never complains about pain - so this must be bad. After he has been seen by the doctor, the appendix appears to be the problem and the boy needs to have it removed. Dad wants his son's pain to go away but is worried because he once got a high dose of a medication and had some unwanted side effects.

Hospital Scene #2: A 14-year-old girl has been experiencing migraine headaches for the past months and is awaiting an appointment with a specialist. Today, however, the pain is the worst it's been. Mom has picked her up from school and brought her to MCH not knowing what else to do to help her. The Advil and Tylenol have not improved her pain. She desperately wants the pain to go away but is worried because she read that some pain medicines are used without any studies done to see if they work and if they are safe. (https://www.ottawalife.com/article/most-medications-prescribed-to-children-have-not-been-adequately-studied?c=9).

In both cases, these children need medicine to help their pain. The treating doctors want to give them pain medicine that will 1) be safe and 2) make the pain go away. This is what parents and the child/teenager, and the doctors want too. Some pain medicines like opioids are often used to help with pain in children. Unfortunately, opioids can have bad side effects and can, when used incorrectly or for a long time, be addictive and even dangerous. A better option would be a non-opioid, like Ketorolac, which also helps pain but is safer and has fewer side effects. The information doctors have about how much Ketorolac to give a child, though, is what has been learned from research in adults. Like with any medication, the smallest amount that a child can take while still getting pain relief is best and safest. Why give more medicine and have a higher risk of getting a side effect, if a lower dose will do the trick? This is what the researchers don't know about Ketorolac and what this study aims to find out.

Children 6-17 years old who are reporting bad pain when they are in the Emergency Department or admitted in hospital and who will be getting an intravenous line in their arm will be included in the study. Those who want to participate will understand that the goal of the study is to find out if a smaller amount of medicine improves pain as much as a larger amount. By random chance, like flipping a coin, the child will be placed into a treatment group. The difference between these treatment groups is the amount of Ketorolac they will get. One treatment will be the normal dose that doctors use at MCH, and the other two doses will be smaller. Neither the patient, parent nor doctor will know how much Ketorolac they are getting. Over two hours, the research nurse or assistant will ask the child how much pain they are in. Our research team will also measure how much time it took for the pain to get better, and whether the child had to take any other medicine to help with pain. The research team will also ask families and patients some questions to understand their perceptions of pain control, pain medicines and side effects they know of.

This research is important because it may change the way that doctors treat children with pain, not just at MCH but around the world. The results of this study will be shared with doctors through conferences and scientific papers. It's also important that clinicians share information with parents and children so that they can understand more about pain medicines and how these medicines can be used safely with the lowest chance of side effects.

DETAILED DESCRIPTION:
Comparison of Ketorolac at Three Doses In Children With Acute Pain: A Randomized Controlled Trial (KETODOSE TRIAL)

Background: Despite the ongoing opioid crisis, opioids remain a commonly prescribed analgesic for patients with acute pain. Ketorolac is the leading parenteral non-steroidal anti-inflammatory drug (NSAID) in Canada commonly used in the Emergency Department (ED) and inpatient settings for acute abdominal pain and migraine headaches. Though it has safer adverse event profile than opioids, its use in children is off label as there are virtually no pediatric trials to inform this practice. Currently the recommended dosing for children is 0.5 mg/kg to a maximum dose of 30 mg. Recent trials with adults have shown no added analgesic benefit to higher doses of ketorolac, when comparing 10 mg to 15 mg or 30 mg, intravenous (IV). A lower dose will be desirable if it achieves similar reduction of pain, as it allows for safer cumulative daily dosing and lower rates of adverse events. This has led many physicians to change their adult practice to a maximum dose of 10 mg IV; however, despite their smaller size, most children continue to be exposed to doses of 30 mg IV, due to a lack of similar available evidence.

Research Question: In children aged 6 - 17 years, with moderate to severe pain (measured using the 11-point verbal numerical rating scale (VNRS)), who are prescribed IV Ketorolac by their treating physician, is low-dose IV Ketorolac (0.25 mg/kg/dose up to 10 mg OR 0.5 mg/kg/dose up to 10 mg) non-inferior (NI) to standard treatment (0.5 mg/kg/dose up to 30 mg) in reducing mean pain scores within a NI margin of 1?

Study Design: Our trial is a single-center, block randomized, double-dummy, double-blind, three-arm, controlled trial with parallel groups. Participants will include: (i) ≥6 years; (ii) with moderate-severe pain (defined as VNRS > 4; (iii) seen in the ED or inpatient setting; and (iv) who have an IV access planned/available. These individuals will be randomized to an arm with active ketorolac and a 'placebo' ketorolac of a differing dose, to maintain blinding through the double-dummy design: (1) standard-dose ketorolac (0.5 mg/kg IV up to 30 mg IV) + low-dose ketorolac placebo; (2) low-dose ketorolac (0.25 mg/kg up IV up to 10 mg IV) + standard-dose ketorolac placebo; or (3) low-dose ketorolac (0.5 mg/kg IV up to 10 mg) + standard-dose ketorolac placebo.

Participants will be allowed any other non-NSAID rescue therapy at any point after our trial drugs are administered, based on clinical team discretion. Based on available adult literature, a chosen NI margin of 1 point (50% of the established MID), an expected mean difference of 0.2 on the VNRS, and standard deviation of 1.5 points, 57 participants will be needed in each group to achieve a 5% alpha at 80% power.

Primary Outcomes: Between each low-dose ketorolac group and standard group mean differences in pain as measured on VNRS at 60 minutes.

Summary: Acute pain requiring parenteral analgesia is very common amongst Canadian children.Despite data in adults and children supporting preferential NSAID use for acute pain, significant gaps in knowledge regarding safe and effective Ketorolac dosing in children still exists. The drug's superior adverse effect profile and lack of dependence and abuse potential, makes this an appropriate than opioids, and is not known to be a substance of misuse.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6.0 years to <18 years: primary outcome measure, 11-point vNRS is validated for use in children ≥6 years, and no other evidence-based acute pain measure is recommended for use in younger children Currently experiencing moderate to severe pain (self-reported pain score >4 using the vNRS at the time of enrollment; ketorolac is used to treat moderate to severe pain)
2. Patients seen in the ED or inpatient setting with acute pain ≤30 days in duration
3. Patient with IV cannula in situ or ordered (to minimize any additional pain or distress)

Exclusion Criteria:

1. Previous enrollment in trial (to ensure all observations are independent and not paired)
2. Post-operative patient (as this included medically induced pain, versus pathology-only)
3. Ketorolac 6 hours and/or opioids 4 hours prior to recruitment (avoid over-dosing and confounding)
4. Use of daily analgesic for any indications (confounding as response to analgesics maybe altered)
5. Caregiver and/or child cognitive impairment (precludes the ability to respond to study questions)
6. History of gastrointestinal bleed or ulcers, inflammatory bowel disease, coagulation disorders, cerebrovascular bleeding, known arterio-vascular malformations (increased bleeding risk)
7. History of chronic and active renal disease, excluding renal calculi and urinary tract infections
8. History of chronic and active hepatocellular disease (ketorolac is metabolized in the liver)
9. Known pregnancy at the time of enrollment (risk of closure of patent ductus arteriosus in fetus)
10. Known hypersensitivity to NSAIDs or opioids
11. Inability to obtain consent (language barrier and the absence of language translator)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Pain relief | 60 minutes post drug administration
  Between each low-dose ketorolac group (B1 and B2) and standard group (A) mean differences in pain as measured on an 11-point verbal Numerical Rating Scale (0 is no pain and 10 is worst pain ever)

SECONDARY OUTCOMES:
Pain relief | 8 hours post study drug administration
  11-point verbal Numerical Rating Scale (0 is no pain and 10 is worst pain ever) score at 30, 90 and 120 minutes as well as 6 to 8 hours post administration.
Pain relief by a minimally important difference (MID) | 60 and 120 minutes post study drug administration
  Proportion of participants who achieves the 2-point reduction in the 11-point verbal numerical rating scale MID pain score reduction.
Change in category of pain | 30, 90, 120 minutes and 6 hours post study drug administration
  Proportion of participants who change the severity of their baseline pain category at all time points (mild = 0 to 3, moderate = 4 to 6, severe ≥7 on the verbal numerical rating scale)
Time to effective analgesia | Within 8 hours post study drug administration
  time at which a verbal numerical rating scale <3 is achieved post-intervention
Rescue analgesia use | Within 8 hours post study drug administration
  Proportion of participants requiring rescue analgesia in each trial arm
Opioid sparing | Within 8 hours post study drug administration
  The total amount of opioids administered as measured by morphine equivalent mg/kg

OTHER OUTCOMES:
Safety outcome 1 | Within 8 hours post study drug administration
  The proportion of children experiencing any adverse events (AEs), as reported by caregivers or clinical staff, will be recorded in accordance with the CONSORT Harms checklist. We will solicit specific expected AEs that are commonly reported with NSAIDs such as gastric pain. Additionally, we will have open-ended questions to collect information on any additional unexpected AEs.
Safety outcome 2 | Within 8 hours post study drug administration
  Frequency of each specific AE (e.g., nausea, vomiting)
Survey to understand patients' and caregivers' knowledge, attitudes, perceptions, and emotions on pain, medications, and their use in treating acute pain. | Within 7-days of pain outcome completion.
  Semi-structured survey with baseline demographics, closed-ended questions (7-point Likert scale)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - McMaster Children's Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared to individual researchers with reasonable request made to the primary investigator and within what is permitted by Hamilton integrated Review Ethics Board.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 20 years

REFERENCES:
- [Derived] Eltorki M, Carciumaru R, Ali S, Holbrook A, Livingston M, Samiee-Zafarghandy S, Beattie K, Thabane L, Giglia L. Comparison of Ketorolac at 3 Doses in Children With Acute Pain: Protocol for A Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 26;14:e76554. doi: 10.2196/76554. PMID 41066173